CLINICAL TRIAL: NCT03159754
Title: Optimal Care of Complicated Appendicitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Steven W. Bruch, Associate Professor of Surgery, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00103791
Record Dates: First submitted 2017-05-17; First posted 2017-05-19 (Actual); Results first posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Appendicitis; Perforated Appendicitis; Ruptured Appendicitis; Complicated Appendicitis
MeSH Terms: conditions — Appendicitis | interventions — Anti-Bacterial Agents; Piperacillin, Tazobactam Drug Combination; Piperacillin; Tazobactam; Ciprofloxacin; Metronidazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Early Appendectomy (Experimental)
  Interventions: Procedure: Early Appendectomy; Drug: Antibiotics
- Interval Appendectomy (Experimental)
  Interventions: Procedure: Interval Appendectomy; Drug: Antibiotics
- No Appendectomy (Experimental)
  Interventions: Drug: Antibiotics

INTERVENTIONS:
Procedure: Early Appendectomy — Removal of the appendix within 24 hours of admission
  Arms: Early Appendectomy
Procedure: Interval Appendectomy — Removal of the appendix after initial antibiotic treatment and at least 6 weeks of recovery.
  Arms: Interval Appendectomy
Drug: Antibiotics — Zosyn will be administered unless the patient has a penicillin allergy, in which case patients will receive both ciprofloxacin and metronidazole.
  Other Names: Zosyn (piperacillin/tazobactam); ciprofloxacin; metronidazole

SUMMARY:
When the appendix becomes infected and inflamed, it is called appendicitis. Sometimes, if the infection and inflammation get worse, the appendix can die or burst, leading to a larger infection or even pus pockets around the appendix. This is called complicated, or perforated, appendicitis. Three common treatments for complicated appendicitis are

* appendectomy (removal of the appendix) right away
* appendectomy several weeks after the diagnosis
* treating the appendicitis without performing an appendectomy

This study seeks to determine which of these three approaches is most cost-effective in children with complicated appendicitis.

DETAILED DESCRIPTION:
This is a single center, prospective study to compare early appendectomy vs. non-operative management of immunocompetent patients with complicated appendicitis, and then to compare interval appendectomy vs. no interval appendectomy in those managed with the initial non-operative approach. Patients who choose early appendectomy will have surgery within 24 hours of diagnosis and be discharged once they are afebrile for 24 hours, have a normal WBC count, and can tolerate a diet. They will be discharged with 5 days of oral ciprofloxacin and metronidazole and follow-up in clinic 2-4 weeks later. Patients who choose non-operative management will receive piperacillin-tazobactam with or without abscess drainage until they are afebrile 24 hours with a normal WBC count and are tolerating a diet, followed by 5 days of oral ciprofloxacin and metronidazole upon discharge. These patients will then be seen in clinic in 2-4 weeks, at which time they will be given the choice of whether or not to undergo interval appendectomy at least 8 weeks from initial presentation. Those in the interval appendectomy group will follow-up one month post-operatively. Patients in both groups will be contacted 3 months and 2 years following initial presentation.

{{{While 40 participants were enrolled as intended, and some data was collected from them, a combination of staff turnover and subsequent resource constraints did not permit the analysis originally intended. Thus, results data is shown comparing the early appendectomy participants against the other two arms combined.}}}}

ELIGIBILITY:
Inclusion criteria

1. At least 1 of the following CT or MRI findings:

   1. Peri-appendicular abscess
   2. Extruded appendicolith
   3. Visible hole in appendiceal wall
   4. Free peritoneal air

   OR
2. CT or MRI read with phlegmon or diffuse/extensive inflammation/free fluid plus 1 of 3 of the following (with CT) or 2 of 3 of the following (with MRI) *:

   1. White blood cell count (WBC) >15
   2. Peritonitis (involuntary right lower quadrant (RLQ) guarding, + Rovsing sign, percussion tenderness, and/or rebound tenderness)
   3. Temperature > 38.0 C *>90% specificity for complicated appendicitis based on unpublished institutional data

Exclusion Criteria

1. Immunocompromized state
2. History of major abdominal operation
3. Previous appendicitis
4. Major comorbidities that preclude safe operation
5. Inability to follow-up or appropriately consent
6. Pregnant women
7. Allergy to penicillin plus any one of the following:

   1. Hypersensitivity to ciprofloxacin and/or metronidazole
   2. Pregnant/lactating women
   3. Patients taking theophylline
   4. Patient taking tizanidine

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven W. Bruch, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Early Appendectomy | Interval Appendectomy | No Appendectomy
Started | 24 | 12 | 4
Completed | 23 | 12 | 4
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Appendectomy | Interval Appendectomy | No Appendectomy | Total
Number analyzed (Participants) | 24 | 12 | 4 | 40
Age, Customized [Count of Participants; unit: Participants]
  5-7 years | 4 | 6 | 2 | 12
  8-12 years | 11 | 5 | 1 | 17
  13-17 years | 9 | 1 | 1 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 0 | 12
  Male | 15 | 9 | 4 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 3
  Not Hispanic or Latino | 21 | 11 | 4 | 36
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: one participant in Early Appendectomy self-identified as "other", rather than any of the NIH/OMB categories
  Participants
    Other: number analyzed (Participants) | 23 | 12 | 4 | 39
    Other: American Indian or Alaska Native | 2 | 0 | 0 | 2
    Other: Asian | 0 | 0 | 1 | 1
    Other: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Other: Black or African American | 0 | 0 | 0 | 0
    Other: White | 20 | 12 | 3 | 35
    Other: More than one race | 0 | 0 | 0 | 0
    Other: Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 12 | 4 | 40

OUTCOME MEASURES:

1. Primary Outcome: Overall Cost of Care
Description: Total health care cost starting from time of admission was the intention of this outcome measure. However, the institutions potentially involved were unwilling to provide access to any cost data so this could not be analyzed for any length of time.
Time Frame: The original intention was to gather cost data for 2 years per person following admission. As no cost data was able to be procured, there is no time frame to which it applies.
Population: No cost data for any participants was able to be procured. Thus this outcome could not be achieved or analyzed in any fashion.
Arm/Group | Early Appendectomy | Interval Appendectomy | No Appendectomy
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Complications
Description: Number of persons who experience any of a number of specified complications, including new/recurrent abscess, wound infection, small bowel obstruction, or need for a larger operation
Time Frame: During index/initial hospitalization (generally not more than 5-6 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Early Appendectomy | Interval Appendectomy | No Appendectomy
Number analyzed (Participants) | 24 | 12 | 4
Participants | 9 | 6 | 1

3. Secondary Outcome: Parents Away From Work
Description: Parents away from work measured in days is presented here. The intention was to collect "missed activity days" for children as well as missed parent work days. However, the question to capture this information referred to school and was determined to be too inconsistent with the way the question may have been interpreted when the survey was given to code reliably.
Time Frame: During index/initial hospitalization (generally not more than 5-6 weeks)
Population: Data shown is all that is available - multiple individuals' data is not available.
Measure: Mean (Full Range); unit: days
Arm/Group | Early Appendectomy | Interval Appendectomy | No Appendectomy
Number analyzed (Participants) | 11 | 4 | 2
days | 7.6 [1 to 21] | 9.3 [1 to 16] | 3.5 [3 to 4]

4. Secondary Outcome: Duration of Antibiotic Therapy
Description: Duration of antibiotic therapy measured in days
Time Frame: During index/initial hospitalization (generally not more than 5-6 weeks)
Population: One person's data from the early appendectomy and four persons from the interval appendectomy for this outcome measure is unavailable.
Measure: Mean (Full Range); unit: days
Arm/Group | Early Appendectomy | Interval Appendectomy | No Appendectomy
Number analyzed (Participants) | 23 | 8 | 4
days | 6.3 [5 to 17] | 5.1 [2 to 6] | 5.4 [5 to 10]

5. Secondary Outcome: Length of Stay
Description: Length of all hospital stays measured in days
Time Frame: During index/initial hospitalization (generally not more than 5-6 weeks)
Measure: Mean (Full Range); unit: days
Arm/Group | Early Appendectomy | Interval Appendectomy | No Appendectomy
Number analyzed (Participants) | 24 | 12 | 4
days | 7.8 [0 to 26] | 7.4 [2 to 32] | 3.5 [2 to 5]

6. Secondary Outcome: Number of Percutaneous Drainage Procedures
Description: Number of persons with differing numbers of percutaneous drainage procedures
Time Frame: During index/initial hospitalization (generally not more than 5-6 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Early Appendectomy | Interval Appendectomy | No Appendectomy
Number analyzed (Participants) | 24 | 12 | 4
Participants
  1 drainage | 4 | 4 | 1
  2 drainage procedures | 1 | 0 | 0

7. Secondary Outcome: Number of Radiographic Imaging Studies
Description: Number of radiographic imaging studies including ultrasound, CT, and MRI
Time Frame: During index/initial hospitalization (generally not more than 5-6 weeks)
Measure: Mean (Full Range); unit: number of imaging procedures/participant
Arm/Group | Early Appendectomy | Interval Appendectomy | No Appendectomy
Number analyzed (Participants) | 24 | 12 | 4
number of imaging procedures/participant | 1.96 [1 to 6] | 2.04 [1 to 6] | 1.88 [1 to 5]

8. Secondary Outcome: Quality of Life (PedsQL)
Description: Original QOL outcome measure listed was: Quality of life measured by PedsQL 2 years following discharge. Two year data collected was insufficient to allow for any analysis. One month GI QOL data collected, also listed in the protocol, is shown below. GI QoL is a validated measure with scores ranging from 0 to 100, where lower scores mean worse quality of life and higher scores mean better quality of life. Peds QL is a validated measure with scores ranging from 0 to 100, where lower scores mean worse quality of life and higher scores mean better quality of life.
Time Frame: 1 month; for GI QOL; 2 years for Peds QL
Population: population sizes listed represent the full number of surveys collected for 1 month GI QOL; For 2 year Peds QL, only one participant provided data for the Interval and No Appendectomy arms, so it is not shown to preserve confidentiality; similarly for early appendectomy, there was only 1 child (as opposed to teens) who completed the survey, so it is not included either.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Early Appendectomy | Interval Appendectomy | No Appendectomy
Number analyzed (Participants) | 17 | 7 | 4
score on a scale
  1 month GI QOL | 80.18 [61 to 100] | 88.4 [79 to 94] | 87.25 [76 to 97]
  2 year Peds QL (parental report): number analyzed (Participants) | 3 | 0 | 0
  2 year Peds QL (parental report) | 86.3 [59.69 to 100] |  |
  2 year Peds QL teen report: number analyzed (Participants) | 3 | 0 | 0
  2 year Peds QL teen report | 87.34 [62.81 to 100] |  |

9. Secondary Outcome: Recurrent Appendicitis
Description: Number of persons who experience recurrent appendicitis requiring hospitalization. Because the early appendectomy arm participant by definition have no appendix to infect after surgery, they are not shown below.
Time Frame: 2 years; (Although this appears longer than trial duration, study completion date is based on last 2 year survey turned in, and medical record analysis looked a full two years per participant which extended a bit longer.)
Measure: Count of Participants; unit: Participants
Arm/Group | Interval Appendectomy | No Appendectomy
Number analyzed (Participants) | 12 | 4
Participants | 2 | 0

ADVERSE EVENTS:
Time Frame: Three months
Description: Participants were followed systematically for 3 months; and records review occurred at 2 years solely for the purpose of readmission for appendicitis (as shown in Outcome Measure 9) so that line of AE data (recurrent appendicitis) alone represents 2 year data.
Arm/Group | Early Appendectomy | Interval Appendectomy | No Appendectomy
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/12 | 0/4
Serious Adverse Events (participants affected / at risk) | 3/24 | 2/12 | 0/4
Other Adverse Events (participants affected / at risk) | 10/24 | 5/12 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Early Appendectomy (N=24) | Interval Appendectomy (N=12) | No Appendectomy (N=4)
Admission for C-Diff (Gastrointestinal disorders) | 1 | 0 | 0
Testicular Swelling-hydrocele (Reproductive system and breast disorders) | 1 | 0 | 0
ED Admission - Fever and Abdominal Pain (General disorders) | 1 | 0 | 0
Recurrence of Appendicitis (Gastrointestinal disorders) | 0 | 2 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Early Appendectomy (N=24) | Interval Appendectomy (N=12) | No Appendectomy (N=4)
Abscess and Drain Placement (Surgical and medical procedures) | 4 | 4 | 1
Abscess (Infections and infestations) | 0 | 1 | 0
Drain Placement (Surgical and medical procedures) | 3 | 0 | 0
Nausea and vomiting (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal Pain (General disorders) | 1 | 0 | 1
Headache (General disorders) | 1 | 0 | 0
Persistent Abscess (Infections and infestations) | 1 | 0 | 0
Redness and discomfort around drain exit site (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Abscess, drainage without drain placement (Infections and infestations) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-05): https://cdn.clinicaltrials.gov/large-docs/54/NCT03159754/Prot_SAP_000.pdf